CLINICAL TRIAL: NCT05002790
Title: A Magnetic Resonance Imaging Study of Changes in the Angle Between the Tracheal and Laryngeal Axes in the Sniffing, Neutral and Extended Head and Neck Positions for Videolaryngoscopy
Brief Title: An MRI Study of the Sniffing, Neutral and Extended Head and Neck Positions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 282078
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-06

CONDITIONS: Intubation, Intratracheal
Keywords: Airway management; Videolaryngoscopy; Hyperangulated blades

STUDY DESIGN:
Intervention Model Description: Single group assignment Controlled trial without randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Data collection (Experimental): All 20 anticipated subjects to be scanned under MRI, with data collected and analysed together
  Interventions: Diagnostic Test: Data collection group

INTERVENTIONS:
Diagnostic Test: Data collection group — Magnetic resonance imaging (MRI) allows measurement of the axes described to suggest which head and neck position would provide best anatomical alignment to reduce anterior impingement.
  All the MRI scans will be conducted using 3.0 Tesla (Optima 750w, GE Medical, Milwaukee, WI, USA) using the cervical spine section of the coil. T2-weighted images in the sagittal plane will be acquired using a fast recovery fast spin echo (FRFSE) technique. The scans will take around two and half minutes and a member of the anaesthetic investigator team will be present to facilitate positional changes and maintain consistency. MRI scanning will be performed in following 3 head and neck positions:
  Neutral position, Sniffing position and the Extension position.

SUMMARY:
The traditional method of tracheal intubation requires the insertion of a laryngoscope into the oral cavity and directly visualisation of the glottis. The traditional head position called the sniffing the morning air position; consisting of lower cervical flexion and extension of the atlanto-occipital joint is commonly used to facilitate tracheal intubation in this manner by aligning the oral axes and providing the operator a view of the glottis.

With the advancement of technology, has seen videolaryngoscopes (VL) developed to ease tracheal intubation. With VL, the glottis is seen through a camera connected to a viewing screen either attached to the top of the laryngoscope or connected to a camera screen by cable. One of the main drawbacks with VL is that a good view of the glottis is seen on the screen, but it can be difficult to pass the tracheal tube through the glottis in comparison to the traditional intubation technique described above. One of the main factors the authors suggest is that VL-assisted intubation requires a head and neck position that is different to the sniffing the morning air position.

This study aims to assess the oral axes in three different head and neck positions under MRI to assess which positions improve axial alignment the most.

DETAILED DESCRIPTION:
The traditional method of tracheal intubation requires the insertion of a laryngoscope with the left hand into the oral cavity to displace the tongue and directly visualise the glottis.

The sniffing the morning air (or sniffing) position has been traditionally used for tracheal intubation using direct laryngoscopy. This comprises of flexion of the lower cervical spine, extension at the atlanto-occiptal joint and a horizontal level between the tragus of the ear and sternum. The theoretical purpose of this position is to improve the glottic visualisation by aligning the oral, pharyngeal and tracheal axes.

In recent years with the advancement of technology, videolaryngoscopy has become popular and many centres are now using only videolaryngoscopes for tracheal intubation. Visualisation occurs indirectly through fibreoptic or digital channels. Most videolaryngoscopes use two types of blades. The Macintosh type for normal airway and hyper-angulated blade for difficult airway.

Hyperangulated blades such as the Glidescope LoPro (Verathon Inc, Bothwell, WA, USA), McGrath Series 5 X blade (Medtronic, Minneapolis, MN, USA) and Storz C-Mac D-blade (Karl Storz Endoscoke, Tuttlingen, Germany) are more curved than the traditional standard geometry used with direct laryngoscopy and are thought to improve glottis visualisation without significant change in head position. However, visualisation of glottis is one of the three steps involved in videolaryngoscopy assisted tracheal intubation. The other two steps include aligning the tube with the glottic inlet and advancing the tube through the glottis into the trachea.

One of the main drawbacks in videolaryngoscopy is that despite good view of glottis on the screen, it can be difficult to successfully advance the tracheal tube into the trachea. Anterior impingement of the tracheal tube at the sub-glottic region is a recognised problem with hyperangulated and channelled videolaryngoscopes. VL directs the pre-formed tracheal tube anteriorly but the trachea descends posteriorly into the thorax creating an acute angle impeding passage of the tube. This can result in difficult intubation or a failed intubation. Manoeuvres such as tube rotation and rotation of bougie can rectify this problem to some extent.

A previous study found that laryngoscopy was more difficult with hyper-angulated blades in the sniffing position as compared to neutral position, contradictory to traditional laryngoscopy teaching. Intermediary positions between sniffing and supine should be studied as these may balance the needs of maintaining sufficient mouth opening and not hindering angles affecting the axial alignment. Both studies recommend the benefits of a ramped position as it does reduce the time to desaturation and reduces aspiration risk compared to supine neutral positions and should be considered when using hyperangulated blades. .

Using magnetic resonance imaging in awake and healthy patients, Adnet, et al. measured the oral, pharyngeal and tracheal axes using the neutral position, sniffing position and simple head extension and found neither position resulted in perfect alignment of the 3 axes. However, they did not study the effect of position on angle between tracheal and laryngeal axes. The search for further evidence is necessary for VL as there is a paucity of research in with regard to best head and neck position for videolaryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent
* Volunteers, UHCW staff, aged > 18 years
* Medically able and willing undertake MRI scanning.
* Should pass the MRI safety check list to enter the MRI suite. All participants will complete an MR safety questionnaire immediately prior to their MR scan

Exclusion Criteria:

* Unable to provide consent
* Not willing to have MRI scan or unable to undergo MRI scanning
* Known difficult intubation, Restricted or neck extension not possible or presence of arthritis of cervical spine.
* For MRI safety reasons all participants with a cardiac pacemaker or other electronic implants will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abramson ZR, Susarla S, Tagoni JR, Kaban L. Three-dimensional computed tomographic analysis of airway anatomy. J Oral Maxillofac Surg. 2010 Feb;68(2):363-71. doi: 10.1016/j.joms.2009.09.086. Epub 2010 Jan 15. PMID 20116709
- [Background] Adnet F, Borron SW, Dumas JL, Lapostolle F, Cupa M, Lapandry C. Study of the "sniffing position" by magnetic resonance imaging. Anesthesiology. 2001 Jan;94(1):83-6. doi: 10.1097/00000542-200101000-00017. PMID 11135726
- [Background] Adnet F, Baillard C, Borron SW, Denantes C, Lefebvre L, Galinski M, Martinez C, Cupa M, Lapostolle F. Randomized study comparing the "sniffing position" with simple head extension for laryngoscopic view in elective surgery patients. Anesthesiology. 2001 Oct;95(4):836-41. doi: 10.1097/00000542-200110000-00009. PMID 11605921
- [Background] Aziz MF, Bayman EO, Van Tienderen MM, Todd MM; StAGE Investigator Group; Brambrink AM. Predictors of difficult videolaryngoscopy with GlideScope(R) or C-MAC(R) with D-blade: secondary analysis from a large comparative videolaryngoscopy trial. Br J Anaesth. 2016 Jul;117(1):118-23. doi: 10.1093/bja/aew128. PMID 27317711
- [Background] Brindley PG, Simmonds MR, Needham CJ, Simmonds KA. Teaching airway management to novices: a simulator manikin study comparing the 'sniffing position' and 'win with the chin' analogies. Br J Anaesth. 2010 Apr;104(4):496-500. doi: 10.1093/bja/aeq020. Epub 2010 Feb 18. PMID 20167582
- [Background] Cooper RM, Pacey JA, Bishop MJ, McCluskey SA. Early clinical experience with a new videolaryngoscope (GlideScope) in 728 patients. Can J Anaesth. 2005 Feb;52(2):191-8. doi: 10.1007/BF03027728. PMID 15684262
- [Background] El-Orbany M, Woehlck H, Salem MR. Head and neck position for direct laryngoscopy. Anesth Analg. 2011 Jul;113(1):103-9. doi: 10.1213/ANE.0b013e31821c7e9c. Epub 2011 May 19. PMID 21596871
- [Background] Horton WA, Fahy L, Charters P. Defining a standard intubating position using "angle finder". Br J Anaesth. 1989 Jan;62(1):6-12. doi: 10.1093/bja/62.1.6. PMID 2917111
- [Background] Greenland KB, Edwards MJ, Hutton NJ. External auditory meatus-sternal notch relationship in adults in the sniffing position: a magnetic resonance imaging study. Br J Anaesth. 2010 Feb;104(2):268-9. doi: 10.1093/bja/aep390. No abstract available. PMID 20086071
- [Background] Greenland KB, Edwards MJ, Hutton NJ, Challis VJ, Irwin MG, Sleigh JW. Changes in airway configuration with different head and neck positions using magnetic resonance imaging of normal airways: a new concept with possible clinical applications. Br J Anaesth. 2010 Nov;105(5):683-90. doi: 10.1093/bja/aeq239. Epub 2010 Sep 15. PMID 20846964
- [Background] Levitan RM, Heitz JW, Sweeney M, Cooper RM. The complexities of tracheal intubation with direct laryngoscopy and alternative intubation devices. Ann Emerg Med. 2011 Mar;57(3):240-7. doi: 10.1016/j.annemergmed.2010.05.035. Epub 2010 Jul 31. PMID 20674088
- [Background] Meisami T, Musa M, Keller MA, Cooper R, Clokie CM, Sandor GK. Magnetic resonance imaging assessment of airway status after orthognathic surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Apr;103(4):458-63. doi: 10.1016/j.tripleo.2006.07.006. Epub 2006 Oct 27. PMID 17395062
- [Background] Mendonca C, Ungureanu N, Nowicka A, Kumar P. A randomised clinical trial comparing the 'sniffing' and neutral position using channelled (KingVision(R) ) and non-channelled (C-MAC(R) ) videolaryngoscopes. Anaesthesia. 2018 Jul;73(7):847-855. doi: 10.1111/anae.14289. Epub 2018 Apr 16. PMID 29660807
- [Background] Stuck BA, Kopke J, Maurer JT, Verse T, Kuciak G, Duber C, Hormann K. Evaluating the upper airway with standardized magnetic resonance imaging. Laryngoscope. 2002 Mar;112(3):552-8. doi: 10.1097/00005537-200203000-00026. PMID 12148870

RESULTS

PARTICIPANT FLOW:
Groups:
- Data Collection: All 20 anticipated subjects to be scanned under MRI, with data collected and analysed together
  Data collection group: Magnetic resonance imaging (MRI) allows measurement of the axes described to suggest which head and neck position would provide best anatomical alignment to reduce anterior impingement.
  All the MRI scans will be conducted using 3.0 Tesla (Optima 750w, GE Medical, Milwaukee, WI, USA) using the cervical spine section of the coil. T2-weighted images in the sagittal plane will be acquired using a fast recovery fast spin echo (FRFSE) technique. The scans will take around two and half minutes and a member of the anaesthetic investigator team will be present to facilitate positional changes and maintain consistency. MRI scanning will be performed in following 3 head and neck positions:
  Neutral position, Sniffing position and the Extension position.
Period: Overall Study
Arm/Group | Data Collection
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Data Collection
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Angle A Measured on MRI
Description: To determine which patient head and neck positioning significantly improves the angle A. It is defined as the angle between the tracheal axis (TA) and laryngeal axis (LA)
Time Frame: Each subject will undergo 3 MRI scans. Angle A will be measured on each scan at the end of all the scans performed that day. The angles will be measured by 2 investigators.
Population: data from all participants was analysed
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Neutral Position: participants positioned in neutral position
- Sniffing Position: participants position din sniffing position
- Extended Position: participants positioned in extended position
Arm/Group | Neutral Position | Sniffing Position | Extended Position
Number analyzed (Participants) | 20 | 20 | 20
degree | 20.7 (6.8) | 10.8 (6.9) | 30.0 (5.2)

2. Secondary Outcome: Angle B, C, D and E Measured Using MRI
Description: The tracheal axis (TA) is defined as a line passing through the centre of intrathoracic part of trachea to the centre of cricoid cartilage. The laryngeal axes (LA) is defined as a line passing through the centre of cricoid cartilage to the base of the epiglottis. The pharyngeal axis (PA) is defined as a line passing through the anterior portion of the atlas and vertebrae C2. The oral axis (OA) is defined as straight line drawn parallel to the hard palate. The line of vision (LV) is defined as the straight line passing through the inferior extremity of the superior incisors and posterior extremity of the superior portion of the cricoid.
  Angle B is angle between the laryngeal axes (LA) and pharyngeal axes (LA) Angle C is angle between pharyngeal axes (PA) and oral axes (OA) Angle D angle between laryngeal axes (LA) and line of vision (LV) Angle E angle between line of vision (LV) and pharyngeal axes (PA)
Time Frame: Each subject will undergo 3 MRI scans. The angles will be measured on each scan at the end of the scanning performed that day. The angles will be measured by 2 investigators.
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Sniffing Position: participants positioned in sniffing position
Arm/Group | Neutral Position | Sniffing Position | Extended Position
Number analyzed (Participants) | 20 | 20 | 20
degree
  Angle B | 13.0 (6.7) | 17.0 (7.4) | 23.9 (6.5)
  Angle C | 87.8 (6.4) | 69.5 (7.2) | 81.7 (6.0)
  Angle D | 38.8 (6.7) | 27.0 (3.9) | 24.5 (5.3)
  Angle E | 51.3 (5.7) | 43.8 (6.0) | 48.4 (5.0)

ADVERSE EVENTS:
Time Frame: 10 minutes
Arm/Group | Data Collection
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT05002790/Prot_SAP_000.pdf